CLINICAL TRIAL: NCT04761835
Title: Subthreshold Peanut in Infants - Understanding Plasticity
Brief Title: STEP-IT-UP - Peanut Allergy Study for Infants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn in IRB
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00279285
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-03

CONDITIONS: Peanut Allergy; Food Allergy
Keywords: infant food allergy; treatment study; peanut allergy treatment; increase threshold of peanut intake for peanut allergic children
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Open label, randomized trial (1:1) to either dietary peanut intake or strict avoidance prior to a double blind placebo controlled food challenge 52 weeks later.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dietary Peanut (Active Comparator): Participants in this group will be asked to continue peanut in their diet for 1 year at a dose determined from the double blind placebo controlled food challenge at baseline. After the 1 year period, participants will be given another double blind placebo controlled food challenge which will be used to determine their current peanut threshold. The current peanut threshold will be used to determine which participants will go into clinical care and which will get sustained unresponsiveness food challenges to peanut.
  Interventions: Biological: Peanut powder or peanut butter
- Strict avoidance (No Intervention): Participants in this group will be asked to strictly avoid any peanut in their diet for 1 year. After the 1 year period, participants will be given another double blind placebo controlled food challenge which will be used to determine whether they will transition to daily dietary peanut or continue with clinical care.

INTERVENTIONS:
Biological: Peanut powder or peanut butter — Commercially available peanut powder or peanut butter.
  Arms: Dietary Peanut

SUMMARY:
Multicenter randomized (1:1) trial of strict avoidance versus sub-threshold dietary introduction of peanut in peanut allergic infants 4-14 months of age who react at a minimum cumulative dose of at least 430 mg of peanut protein at initial oral food challenge (OFC) for 12 months, followed by cross-over to sub-threshold dietary introduction of peanut in those randomized initially to avoidance.

ELIGIBILITY:
Inclusion Criteria:

* Children age 4-14 months suspected to be peanut allergic

Exclusion Criteria:

* Significant medical problems

Ages: 4 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Oral food challenge threshold to peanut at week 52 | 52 weeks
  compare the oral food challenge threshold (in milligrams) to peanut during a double-blind placebo-controlled food challenge (DBPCFC) after 12 months between subjects randomized to dietary peanut introduction and those randomized to avoidance.

SECONDARY OUTCOMES:
1. Oral food challenge threshold to peanut at week 52 for those initially randomized to dietary peanut compared to the oral food challenge threshold at week 104 for those initially randomized to strict avoidance | 104 weeks
  Compare the oral food challenge threshold (in milligrams) to peanut during a double-blind placebo-controlled food challenge (DBPCFC) after 12 months of dietary peanut between subjects randomized to dietary peanut introduction first and those randomized to avoidance for 52 weeks and subsequent dietary peanut after week 52.
Oral food challenge threshold at 1 month avoidance after 12 months in each treatment group | 56 weeks
  Comparison of OFC threshold (in milligrams) at 1 month of avoidance (sustained unresponsiveness) after 12 months of dietary peanut between those initially randomized to peanut and those randomized to delayed introduction.
Oral food challenge threshold at 2 months avoidance after 12 months in each treatment group | 60 weeks
  Comparison of OFC threshold (in milligrams) at 2 months of avoidance (sustained unresponsiveness) after 12 months of dietary peanut between those initially randomized to peanut and those randomized to delayed introduction.
Safety with dietary introduction of peanut or avoidance | 52 weeks
  Number of participants who have severe (grade 3) anaphylaxis secondary to any DBPCFC or ingestion of the measured dose of peanut.
Rate of discontinuation of dietary peanut | 104 weeks
  Number of participants randomized to dietary peanut who discontinue peanut.
Severity of eczema as assessed by the Scoring Atopic Dermatitis (SCORAD) score | 104 weeks
  Eczema severity as assessed by the SCORAD. The SCORAD has a component for patient measured outcomes and also provider assessment of eczema involvement. It has an overall score range of 0-100, where higher scores signify more severe eczema.
Peanut skin prick test wheal size | 104 weeks
  Average wheal size (millimeters) of peanut skin prick test for participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Keet, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No
No individual participant level data will be shared. Only aggregate data from the study will be shared.